CLINICAL TRIAL: NCT03054909
Title: QUILT-2.021: Randomized Study of Single Course of Intraperitoneal (IP) ALT-803 Followed by Subcutaneous (SQ) Maintenance ALT-803 Versus Subcutaneous (SQ) Maintenance ALT-803 Only After 1st Line Chemotherapy for Advanced Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: IP ALT-803 Followed by SQ ALT-803 for Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS034
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: FIGO Stage III and IV Ovarian Cancer; FIGO Stage III and IV Fallopian Tube Cancer; FIGO Stage III Primary Peritoneal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: ALT-803 subcutaneous only (Experimental)
  Interventions: Biological: ALT-803 Subcutaneous
- Arm 2: ALT-803 intraperitoneal and subcutaneous (Experimental)
  Interventions: Biological: ALT-803 Intraperitoneal

INTERVENTIONS:
Biological: ALT-803 Subcutaneous — Patient receives ALT-803 10 mcg/kg subcutaneous weekly x 4 followed by 4 weeks of no treatment before continuing with treatment courses 2, 3, and 4. Treatment courses 2, 3, and 4 are identical for all patients - ALT-803 10 mcg/kg subcutaneous weekly x 4 with a 4 week rest (4 weeks on/4 weeks off)
  Arms: Arm 1: ALT-803 subcutaneous only
Biological: ALT-803 Intraperitoneal — Patient receives ALT-803 10 mcg/kg intraperitoneal weekly x 4 weeks followed by 4 weeks of no treatment before continuing with treatment courses 2, 3, and 4. Treatment courses 2, 3, and 4 are identical for all patients - ALT-803 10 mcg/kg subcutaneous weekly x 4 with a 4 week rest (4 weeks on/4 weeks off).
  Arms: Arm 2: ALT-803 intraperitoneal and subcutaneous

SUMMARY:
This is a single center, randomized phase II study of an IL-15Rα-Fc super-agonist complex (ALT-803) given as maintenance therapy after the completion of 1st line IV/IP chemotherapy for the treatment of advanced ovarian, fallopian tube, and primary peritoneal cancer.

DETAILED DESCRIPTION:
In this study all patients receive four 8 week cycles of ALT-803 consisting of 4 weekly doses followed by a 4 week rest (no treatment). As it is not known how intraperitoneal (IP) administration (a route of drug administration frequently used for gynecologic cancers) of ALT-803 compares to subcutaneous (SQ) administration, both routes of administration will be tested. The primary objective of this trial is to select one method of delivery for further testing.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of FIGO stage III or grade IV epithelial ovarian, fallopian tube or primary peritoneal carcinoma, has received at least 3 cycles of first line IV/IP cisplatin and paclitaxel chemotherapy and has stable disease or better - refer to Appendix II for FIGO staging system (Note: to be eligible for this study, the patient must receive a minimum of 3 cycles of IP therapy; however, patients may continue on IV only 1st line therapy for additional cycles as long as inclusion criteria 4.1.2 is met)
* Able to begin study therapy within 3 months of final dose of first line chemotherapy
* Functioning intraperitoneal catheter
* ≥ 18 years of age
* GOG performance status ≤ 2 (Appendix II)
* Adequate organ function within 14 days of enrollment defined as:

  * Hematology: hemoglobin ≥ 8 g/dl, absolute neutrophil count (ANC) ≥ 1500/ul, platelets ≥ 50 x 109/L
  * Creatinine: ≤ 2.0 mg/dL
  * Hepatic: SGOT and SGPT ≤ 3 x upper limit of institutional normal (ULN)
* Ability to be off prednisone and other immunosuppressive drugs for at least 3 days prior to and while receiving ALT-803
* Voluntary written consent prior to the performance of any research related procedures

Exclusion Criteria

* Received any investigational agent within the 14 days before the start of ALT-803
* Class II or greater New York Heart Association Functional Classification criteria (Appendix II) or serious cardiac arrhythmias likely to increase the risk of cardiac complications of cytokine therapy (e.g. ventricular tachycardia, frequent ventricular ectopy, or supraventricular tachyarrhythmia requiring chronic therapy)
* Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval greater than 500 milliseconds)
* Uncontrolled bacterial, fungal or viral infections including HIV-1/2 or active hepatitis C/B - chronic asymptomatic viral hepatitis is allowed
* Active autoimmune disease requiring systemic immunosuppressive therapy
* History of severe asthma and currently on chronic systemic medications (mild asthma requiring inhaled steroids only is eligible)
* Uncontrolled hypertension: defined as ≥2 readings over 160 mmHg systolic or 110 mmHg diastolic within month prior to enrollment despite optimal anti-hypertensive medication. Patients with high readings which improve to ≤160/110 after adjustment of medications will be eligible.
* History of pulmonary disease or abnormal pulmonary function studies
* History of narcolepsy or any neurological condition which may impair consciousness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Incidence of Progression Free Survival after first treatment of ALT-803.
Time Frame: 6 months
Population: survival probability estimate
Measure: Number (95% Confidence Interval); unit: Percentage of PFS
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Number analyzed (Participants) | 3 | 4
Percentage of PFS | 50 [1 to 91] | 100 [0 to 100]

2. Secondary Outcome: Progression Free Survival
Description: Incidence of Progression Free Survival after first treatment of ALT-803.. Survival probability estimate.
Time Frame: 1 year
Population: survival probability estimate
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Number analyzed (Participants) | 3 | 4
Percentage of participants | 50 [1 to 91] | 100 [0 to 100]

3. Secondary Outcome: Overall Survival
Description: Overall Survival from start of ALT-803 dosing
Time Frame: 1 year
Population: survival probability estimate
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Number analyzed (Participants) | 3 | 4
Percentage of participants | 100 [0 to 100] | 100 [0 to 100]

4. Secondary Outcome: ALT-803 Associated Toxicities
Description: Incidence of ALT-803 associated toxicities after first treatment of ALT-803.
Time Frame: 1 year
Population: Count of events
Measure: Number; unit: Count of events
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Number analyzed (Participants) | 3 | 4
Count of events | 65 | 100

5. Secondary Outcome: Incidence of Recorded Toxicity Grade 3 or Greater
Description: Grade 3 adverse events or greater will be measured. A Grade 3 adverse event is defined as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling.
Time Frame: 1 year
Population: Count of events
Measure: Number; unit: Number of of adverse events
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Number analyzed (Participants) | 3 | 4
Number of of adverse events | 1 | 2

6. Secondary Outcome: Progression Free Survival
Description: Incidence of Progression Free Survival after first treatment of ALT-803.. Survival probability estimate.
Time Frame: 2 years
Population: survival probability estimate
Measure: Number (95% Confidence Interval); unit: Percentage of PFS
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Number analyzed (Participants) | 3 | 4
Percentage of PFS | 50 [1 to 91] | 100 [0 to 100]

7. Secondary Outcome: Overall Survival
Description: Overall Survival after first treatment of ALT-803.
Time Frame: 2 year
Population: Survival probability estimate
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
Number analyzed (Participants) | 3 | 4
Percentage of participants | 100 [0 to 100] | 100 [0 to 100]

ADVERSE EVENTS:
Time Frame: Patients were monitored from first dose of ALT-803 until two years after off treatment date, 3 years in total.
Arm/Group | Arm 1: ALT-803 Subcutaneous Only | Arm 2: ALT-803 Intraperitoneal and Subcutaneous
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: ALT-803 Subcutaneous Only (N=3) | Arm 2: ALT-803 Intraperitoneal and Subcutaneous (N=4)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: ALT-803 Subcutaneous Only (N=3) | Arm 2: ALT-803 Intraperitoneal and Subcutaneous (N=4)
Injection site reaction (General disorders) | 3 (46) | 4 (48)
Chills (General disorders) | 3 (25) | 4 (12)
Fever (General disorders) | 2 (4) | 3 (5)
Flu like symptoms (General disorders) | 2 (3) | 4 (8)
Pain (General disorders) | 2 (4) | 1 (2)
Gait disturbance (General disorders) | 2 (8) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03054909/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03054909/ICF_001.pdf